CLINICAL TRIAL: NCT04370145
Title: Antibiotics Treatment of Cholangitis Post-Kasai Portoenterostomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Shanghai Children's Hospital (Other)
Responsible Party: Principal Investigator, J.X. Feng, Chief in Department, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JXFeng
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Cholangitis, Secondary Biliary; Treatment Compliance; Antibodies Drug Specific
Keywords: Cholangitis; biliary atresia; kasai Portoenterostomy; antibiotics; treatment
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Patient Compliance; Cholangitis; Biliary Atresia | interventions — sulperazone; Tinidazole; Teicoplanin; Meropenem

STUDY DESIGN:
Intervention Model Description: Cholangitis patients post-kasai Portoenterostomy were grouped by cholangitis severity score, according to the severity was divided into mild, moderate, severe cholangitis, all levels of cholangitis patients were divided into subgroups by age and post-kasai Portoenterostomy jaundice matching design of experiment, then they were randomly divided into control group and experimental group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- moderate cholangitis (Experimental): Meropenem injection, iv. drip,20mg/Kg，Q12h; Tinidazole injection, iv. drip,20mg/Kg,Qd.
  Interventions: Drug: Sulperazon
- severe cholangitis (Experimental): Meropenem injection, iv. drip,20mg/Kg，Q8h; Teicoplanin injection, iv. drip,10mg/Kg,Qd; Tinidazole injection, iv. drip,20mg/Kg,Qd.
  Interventions: Drug: Teicoplanin
- control group (Active Comparator): Sulperazon, iv.,drip,100mg/Kg,Bid; Tinidazole injection, iv. drip,20mg/Kg,Qd
  Interventions: Drug: Meropenem Injection

INTERVENTIONS:
Drug: Sulperazon — moderate cholangitis patients were treated with these drugs for 7days,unless the patients were cured or must be changed the therapeutic.
  Other Names: Tinidazole injection
  Arms: moderate cholangitis
Drug: Teicoplanin — severe cholangitis patients were treated with these drugs for 7days,unless the patients were cured or must be changed the therapeutic.
  Other Names: Meropenem Injection; Tinidazole injection
  Arms: severe cholangitis
Drug: Meropenem Injection — cholangitis in control group were treated with these drugs for 7days,unless the patients were cured or must be changed the therapeutic.
  Other Names: Tinidazole injection
  Arms: control group

SUMMARY:
Application of multi-center, prospective study on the severity of postoperative cholangitis biliary atresia classification, according to the degree of cholangitis targeted therapy, to improve the therapeutic effect of postoperative cholangitis biliary atresia, decrease the overuse of antibiotics related complications.

DETAILED DESCRIPTION:
Cholangitis patients post-kasai Portoenterostomy were grouped by cholangitis severity score, according to the severity was divided into mild, moderate, severe cholangitis, all levels of cholangitis patients were divided into subgroups by age and post-kasai Portoenterostomy jaundice matching design of experiment, then they were randomly divided into control group and experimental group, and all the control group unified antibiotic treatment, the experimental group was graded antibiotic treatment according to the severity cholangitis, after three days treatment，evaluate each treatment effect, average hospitalization days, the average hospitalization expenses, antimicrobial drug use strength to evaluate the therapeutic effect of postoperative cholangitis biliary atresia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 months to 2 years old, gender is not limited.
2. Patients with cholangitis post-kasai Portoenterostomy.
3. No other treatment before entering the group.
4. The patient must sign an informed consent form and can actively cooperate with the treatment and follow-up.

Exclusion Criteria:

1. Patients with other infectious lesions.
2. Patients with other severe deformity.
3. Patients with end-stage liver failure.
4. Patientsn with liver transplantation.
5. Patients with mental symptoms or other disease.

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Recovery rate | 7 days
  The cure indicator including:1.Temperature:T≤37.5℃; 2. Infection index:WBC<10x109/L, CRP<10mg/L. After 7days treatment, we calculate the cure number and recovery rate of each group to evaluate the efficiency.

SECONDARY OUTCOMES:
Recurrence rate | 1 year
  To collect recurrent episode of cholangitis and recurrent rate of each group.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Jiexiong, Postdoctoral, Principal Investigator — Tongji Hospital
Locations (2):
- China (2):
  - Tongji hospital affiliated to tongji medical college of huazhong university of science and technology, Wuhan, Hubei
  - TongjiHospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang P, Zhang HY, Yang J, Zhu T, Wu X, Yi B, Sun X, Wang B, Wang T, Tang W, Xie H, Tou J, Han Y, Liu X, Zhan J, Liu Y, Li Y, Lv Z, Lu L, Zhao B, Fu T, Wu D, Bai J, Li W, Yang H, Zhang G, Ren H, Feng J. Severity assessment to guide empiric antibiotic therapy for cholangitis in children after Kasai portoenterostomy: a multicenter prospective randomized control trial in China. Int J Surg. 2023 Dec 1;109(12):4009-4017. doi: 10.1097/JS9.0000000000000682. PMID 37678274